CLINICAL TRIAL: NCT02770118
Title: Effects of Sleep Restriction on BAT Activation in Humans
Acronym: BAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: New York University (Other)
Responsible Party: Principal Investigator, Marie-Pierre St-Onge, Assistant Professor of Nutritional Medicine, Dept of Medicine Endocrinology, Columbia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AAAQ1008
Record Dates: First submitted 2016-02-10; First posted 2016-05-12 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Sleep Deprivation; Obesity
Keywords: sleep restriction; obesity; brown adipose tissue
MeSH Terms: conditions — Sleep Deprivation; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PSR-TSD (Experimental): Partial sleep restriction (PSR) followed by total sleep deprivation (TSD). Experimental procedures will begin with a 3-day period of habitual sleep (HS).
  Interventions: Behavioral: Partial Sleep Restriction; Behavioral: Total Sleep Deprivation; Behavioral: Habitual Sleep
- TSD-PSR (Experimental): Total sleep deprivation (TSD) followed by partial sleep restriction (PSR). Experimental procedures will begin with a 3-day period of habitual sleep (HS).
  Interventions: Behavioral: Partial Sleep Restriction; Behavioral: Total Sleep Deprivation; Behavioral: Habitual Sleep

INTERVENTIONS:
Behavioral: Partial Sleep Restriction — 4 hour time in bed (TIB), participants will go to bed 4 hours later than during the HS condition. Wake-up times will be the same. During the in-lab portion of the PSR, meals, fulfilling weight-maintenance energy requirements, will be supplied by the research staff as BOOST shakes.
  Other Names: PSR
Behavioral: Total Sleep Deprivation — 0 hour time in bed (TIB), participants will remain awake throughout the night. Meals will be provided as BOOST shakes at the same meal.
  Other Names: TSD
Behavioral: Habitual Sleep — 8 hours time in bed (TIB), for 3 nights, with fixed bed and wake times, while at home. During the 3-d HS phase, participants will be provided will BOOST meal replacement shakes in amounts required to achieve weight maintenance.
  Other Names: HS

SUMMARY:
The goal of this proposed research is to test the hypothesis that long-term mild sleep restriction (SR), as occurs frequently in adults and adolescents, leads to a positive energy balance and weight gain.

Aim 1. To determine the effects of SR, relative to habitual sleep (HS), on food choice and energy intake (EI) in adults at risk of obesity.

* Hypothesis 1a. EI, assessed by multiple weekly 24-hour recalls, will be greater during a period of SR relative to HS. This will be mostly due to increased fat and carbohydrate intakes.
* Hypothesis 1b. Neuronal responses to food stimuli, assessed by functional MRI (fMRI) after 6 weeks of SR or HS, will indicate increased activity in networks associated with reward and food valuation (insula, orbitofrontal cortex) during a period of SR relative to HS. These responses will be correlated with intakes of high carbohydrate and high fat foods (hypothesis 1a) and neuropeptide Y (NPY). Moreover, activation of the default mode network (DMN) will be suppressed to a lesser extent after SR compared to HS.

Aim 2. To determine the effects of SR, relative to HS, on energy expenditure (EE) via independent and complementary approaches.

* Hypothesis 2a. EE, assessed by doubly-labeled water (DLW), and physical activity level, monitored daily by actigraphy, will be lower during SR relative to HS.
* Hypothesis 2b. Brown adipose tissue (BAT), assessed by positron emission tomography and magnetic resonance combined scanner (PET/MR) using 18F-fluorodeoxyglucose (18FDG-PET) and fat fraction (FF) measurement under cold stimulation, will be greater after SR relative to HS. This would suggest higher adaptive thermogenesis after SR compared to HS. BAT activation will also be correlated with NPY.

Aim 3. To determine whether SR alters body weight and adiposity relative to HS.

* Hypothesis 3a. SR will lead to weight gain and increased total adiposity, as assessed using magnetic resonance imaging (MRI), relative to HS.
* Hypothesis 3b. Increased adiposity after SR will be correlated to an adverse cardio-metabolic risk profile (increased glucose, insulin, triglycerides, leptin, reduced high-density lipoprotein cholesterol and adiponectin) and neuronal responses to food stimuli (Hypothesis 1b), and EE (Hypothesis 2a & 2b). Failure to stimulate BAT with SR will be associated with greater gain in adiposity.

DETAILED DESCRIPTION:
There is an association between short sleep duration (SSD) and obesity. Moreover, short sleepers (<7 hours sleep/night) gain more weight over time than normal sleepers (7-8 hours sleep/night). These relationships are increasingly supported by clinical data showing that restricting sleep duration in healthy, normal weight adults, increases energy intake (EI).

ELIGIBILITY:
Inclusion Criteria:

* Normal scores on:

  * Pittsburgh Quality of Sleep Questionnaire
  * Epworth Sleepiness Scale
  * Berlin Questionnaire
  * Sleep Disorders Inventory Questionnaire
  * Beck Depression Inventory
  * Composite Scale of Morningness/Eveningness
  * Three Factor Eating Questionnaire
* Sleep 7-9 hours in bed/night with no daytime nap
* Age 20-49 years, premenopausal women
* All racial/ethnic groups
* Body mass index 25-29.9 kg/m2

Exclusion Criteria:

* Smokers (any cigarettes or ex-smoker <3 years)
* Neurological, medical or psychiatric disorder, diabetics
* Eating and/or sleep disorders
* Contraindications for MRI scanning
* Travel across time zones within 4 weeks
* History of drug and alcohol abuse
* Shift worker (or rotating shift worker)
* Caffeine intake >300 mg/d
* Pregnancy or within 1 y post-partum
* Heavy equipment operators Commercial long-distance drivers

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline Brown adipose tissue (BAT) in 6 weeks | 6 weeks
  Assessed by positron emission tomography and magnetic resonance combined scanner (PET/MR) using 18F-fluorodeoxyglucose (18FDG-PET). Fat fraction (FF) measurement under cold stimulation is to be measured.

SECONDARY OUTCOMES:
Difference in weight from baseline at 6 weeks | 6 weeks
  Assessed by body composition and anthropometric measurements.
Difference in Glucose level from baseline at 6 weeks | 6 weeks
  Assessed by fasting blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, Ph.D, Principal Investigator — Assistant Professor of Nutritional Medicine
Locations (1):
- New York Nutrition Obesity Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No